CLINICAL TRIAL: NCT05062304
Title: Once-Daily Single-Inhaler Triple Versus Dual Therapy in Patients With COPD (IMPACT Trial)
Brief Title: Replication of the IMPACT COPD Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-IMPACT
Record Dates: First submitted 2021-06-21; First posted 2021-09-30 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fluticasone furoate-vilanterol trifenatate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fluticasone furoate-vilanterol: Reference group
  Interventions: Drug: Fluticasone Furoate-Vilanterol Trifenatate
- Fluticasone furoate-umeclidinium-vilanterol: Exposure group
  Interventions: Drug: Furoate-umeclidinium-vilanterol

INTERVENTIONS:
Drug: Fluticasone Furoate-Vilanterol Trifenatate — Fluticasone Furoate-Vilanterol Trifenatate dispensing claim is used as the reference group.
  Groups: Fluticasone furoate-vilanterol
Drug: Furoate-umeclidinium-vilanterol — Furoate-umeclidinium-vilanterol dispensing claim is used as the exposure group.
  Groups: Fluticasone furoate-umeclidinium-vilanterol

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Please see https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

All patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of triple therapy or fluticasone furoate-vilanterol (index date).

Eligible Cohort Entry Dates:

Market availability of fluticasone furoate-umeclidinium-vilanterol in the U.S. for management of COPD was approved by FDA on September 18, 2017.

* For Marketscan: September 18, 2017 - December 31, 2018 (end of available data)
* For Optum: September 18, 2017 - June 30, 2020 (end of available data)

Inclusion Criteria:

* 40 years of age
* Established clinical history of COPD in accordance with the definition by the ATS/ERS
* Receiving daily maintenance treatment for their COPD for at least 3 months prior to screening
* A post-bronchodilator FEV1 < 50% predicted normal and a documented history of ≥ 1 moderate or severe COPD exacerbation in the previous 12 months OR a post-bronchodilator 50% ≤FEV1 < 80% predicted normal and a documented history of ≥ 2 moderate exacerbations or a documented history of ≥1 severe COPD exacerbation (hospitalized) in the previous 12 months.

Exclusion Criteria:

* Pregnancy or child bearing potential without acceptable contraceptive method
* Subjects with α1-antitrypsin deficiency as the underlying cause of COPD
* Subjects with active tuberculosis, lung cancer, significant bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases
* Subjects with lung volume reduction surgery within the 12 months prior to screening
* Immune suppression (e.g. HIV, Lupus) or other risk factors for pneumonia (e.g. neurological disorders affecting control of the upper airway, such as Parkinson's Disease, Myasthenia Gravis)
* Pneumonia and/or moderate or severe COPD exacerbation that has not resolved at least 14 days prior to Screening and at least 30 days following the last dose of oral/systemic corticosteroids (if applicable). In addition, any subject that experiences pneumonia and/or moderate or severe COPD exacerbation during the run-in period will be excluded
* Other Respiratory tract infections that have not resolved at least 7 days prior to screening
* Unstable liver disease as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices or persistent jaundice, cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). Note: Chronic stable hepatitis B and C are acceptable if the subject otherwise meets entry criteria
* Unstable or life threatening cardiac disease: subjects with any of the following at Screening (Visit 1) would be excluded: Myocardial infarction or unstable angina in the last 6 months
* Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months
* NYHA Class IV Heart failure
* Oxygen therapy: Use of long-term oxygen therapy (LTOT) described as resting oxygen therapy >3L/min (Oxygen use less than or equal to 3L/min flow is not exclusionary.)
* Pulmonary rehabilitation: Subjects who have participated in the acute phase of a Pulmonary Rehabilitation Program within 4 weeks prior to Screening or subjects who plan to enter the acute phase of a Pulmonary Rehabilitation Program during the study. Subjects who are in the maintenance phase of a Pulmonary Rehabilitation Program are not excluded
* Drug/alcohol abuse: Subjects with a known or suspected history of alcohol or drug abuse
* The use of any of the following medications under the given conditions:

  * Long term antibiotic use (short term antibiotics are allowed if treating short-term acute infection or short-term exacerbation
  * Use of a systemic, oral, or parenteral corticosteroid in the last 30 days (except unless treating COPD exacerbations/pneumonia)

Ages: 40 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, propensity score-matched, retrospective cohort study design comparing triple therapy to fluticasone furoate-vilanterol users. The patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of triple therapy or fluticasone furoate-vilanterol (index date). We will restrict the analyses to patients with a diagnosis of COPD who have been receiving daily maintenance therapy for at least 3 months prior to index date.
Sampling Method: Non-Probability Sample
Enrollment: 17281 (Actual)
Dates: Start 2020-12-13 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Annual rate of moderate or severe COPD exacerbations during treatment | To study completion or censoring, up to 32 months
  Claims-based algorithm: see attached protocol for full definition

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT05062304/Prot_000.pdf